CLINICAL TRIAL: NCT05155202
Title: Clinical Relevance of Nicardipine Induced Hypoxemia in the Intensive Care Unit. A Multicenter Prospective Observational Study Comparing Nicardipine and Urapidil
Brief Title: Clinical Relevance of Nicardipine Induced Hypoxemia in the Intensive Care Unit
Acronym: ECRHIN-ICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ID2885
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hypoxemic Respiratory Failure; Side Effect; Hypertensive Emergency
MeSH Terms: conditions — Respiratory Insufficiency; Hypertensive Crisis | interventions — Antihypertensive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nicardipine: Major patients hospitalized in intensive care unit, with systolic hypertension, requiring administration of intravenous Nicardipine.
  Interventions: Drug: Antihypertensive Agents
- Urapidil: Major patients hospitalized in intensive care unit, with systolic hypertension, requiring administration of intravenous Urapidil.
  Interventions: Drug: Antihypertensive Agents

INTERVENTIONS:
Drug: Antihypertensive Agents — Administration of intravenous Nicardipine or Urapidil

SUMMARY:
In the context of postoperative hypertension in the intensive care units, or after resusitation of hypertensive patients, intravenous antihypertensive drugs are often used. Among those drugs, Nicardipine is an effective drug, but with side effects such as inhibition of pulmonary vasoconstriction. Only preclinical studies have investigated the pathophysiology of this mechanism, and no clinical study have proven its clinical relevance.

The aim of this study is to establish the incidence of Nicardipine induced hypoxemia and to compare it to another antihypertensive agent, Urapidil.

DETAILED DESCRIPTION:
Prospective observational study in 4 intensive care units in one general hospital and one university hospital.

Once Nicardipine or Urapidil infusion is started, data collection of respiratory related information such as type of ventilation, arterial partial pressure of oxygen, blood pressure, cardiac frequency.

Statistical analysis for two qualitative variables: Group (Nicardipine or Urapidil) and occurrence or worsening of hypoxemia. Secondary outcoumes analysed such as maximal drop of blood pressure, evolution of the PaO2/FiO2 ratio, length of hospital stay, duration of mechanical ventilation in the ventilated patients.

Analysis for different subgroups : Patients with known atelectasis, postoperative of cardiac surgery, neuro-intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* With acute arterial systolic hypertension over 140mmHg
* Requiring intravenous administration of one of the two following drugs : Urapidil or Nicardipine

Exclusion Criteria:

* Patient ventilated Under Nitrogen Monoxyde
* Contraindication to Nicardipine or Urapidil
* Refusal of the patient or his relatives
* Patient treated for pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hypertensive patients in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | During the twelve hours following start of drug infusion
  Occurrence of worsening of hypoxemia

SECONDARY OUTCOMES:
Efficacy of antihypertensive action | During the twelve hours following start of drug infusion
  Time before the drop of arterial systolic blood pressure below 140mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- CHU CAEN, Caen, France

IPD SHARING:
Plan to Share IPD: No